CLINICAL TRIAL: NCT06243562
Title: The Effects Of Progressive Muscle Relaxation Training in Addition to the Combined Exercise Training in Women With Fibromyalgia
Brief Title: The Effects Of Progressive Muscle Relaxation Training in Women With Fibromyalgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Eylem TÜTÜN YÜMİN, Professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIBU-FTR-ETY-03
Record Dates: First submitted 2024-01-23; First posted 2024-02-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; progressive muscle relaxation; combined exercise; rehabilitation
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Intervention Model Description: There will be an intervention and control group in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined exercises and progressive muscle relaxation group (Active Comparator): Participants in this group will be given combined exercises consisting of aerobic exercise, strengthening exercise and stretching exercise, as well as progressive muscle relaxation training. The studies will be carried out under the supervision of a physiotherapist.
  Interventions: Other: combined exercises and progressive muscle relaxation group
- combined exercises group (Active Comparator): Participants in this group will be given combined exercises consisting of aerobic exercise, strengthening exercise and stretching exercise. They will rest for 10-15 minutes in a relaxation position only. The studies will be carried out under the supervision of a physiotherapist.
  Interventions: Other: combined exercises group

INTERVENTIONS:
Other: combined exercises and progressive muscle relaxation group — Participants in the intervention group will receive a combined exercise program that will last 45-60 minutes, 3 days a week for 8 weeks, and progressive muscle relaxation training that will last 10-15 minutes, under the supervision of a therapist.
  Arms: combined exercises and progressive muscle relaxation group
Other: combined exercises group — Patients in the control group will perform a combined exercise consisting of aerobic, strengthening and stretching exercises, which will last 45-60 minutes, 3 days a week for 8 weeks, under the supervision of a physiotherapist. At the end of the combined exercise program, they will rest in the relaxation position for 10-15 minutes each session.
  Arms: combined exercises group

SUMMARY:
The purpose of the study is to examine the effects of progressive muscle relaxation training given in addition to a combined exercise program in women with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia syndrome is a complex, non-inflammatory pain syndrome characterized by whole-body pain, pain at specific tender points, fatigue, and sleep disturbance

The prevalence of fibromyalgia in the world population varies between 0.2% and 6.4%, and it more frequently affects middle-aged women (30-50 years old). the etiology of fibromyalgia is not fully known.

There are no generally accepted objective clinical findings, radiographic abnormalities, or laboratory tests to assess the presence of fibromyalgia and measure fibromyalgia severity. Therefore, questionnaires measuring patients' subjective responses remain important in the evaluation of fibromyalgia patients until now.

Current treatment recommendations for fibromyalgia strongly support a multifaceted regimen, including patient education, physical therapy, massage, cognitive behavioral therapy, specific pharmacotherapy, restorative sleep, and exercise. Exercise includes aerobic exercise, strengthening and stretching.

Progressive muscle relaxation therapy is an alternative complementary therapy based on the principle of progressive tensing and relaxing of major body muscles to relieve psychological tension. The therapy has no time or space restrictions and does not require any special equipment.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with fibromyalgia over the age of 20
* volunteering to participate in the study.

Exclusion Criteria:

* neurological, infectious, endocrine and/or other inflammatory rheumatic diseases
* serious psychiatric illness (schizophrenia, etc.)
* any condition that prevents exercise (advanced heart, respiratory or orthopedic problems)
* Malignancy
* pregnancy
* menopause
* Participating in a physical therapy program (receiving exercise / relaxation training) in the last 6 months

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-04-12 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Eight weeks
  The Visual Analog Scale measures pain intensity. It consists of a 10 cm line with two end points representing 0 (no pain) to 10 (pain as bad as possible). The patient marks the current pain level by placing a mark on the line.
The Pain Catastrophizing Scale | Eight weeks
  The Pain Catastrophizing Scale is a self-report measure of pain-related catastrophizing thinking. It consists of 13 items on a five-point Likert scale (0 = never to 4 = always ). The total score ranges from 0 to 52, with higher scores indicating higher levels of pain catastrophizing.

SECONDARY OUTCOMES:
The Fibromyalgia Impact Scale | Eight weeks
  The Fibromyalgia Impact Scale assesses the severity of fibromyalgia and its impact on daily function. It contains 10 items: subscores are summed to create a scale from 0 to 100, with a higher score indicating worse symptoms and greater dysfunction.
COMPASS 31 Scale: | Eight weeks
  COMPASS 31 scale is a self-assessment tool that investigates autonomic symptoms. The scale contains 31 items assessing six domains of autonomic functions. The total score ranges from 0 (normal) to 100 (worst case).
Skin Temperature | Eight weeks
  Peripheral skin temperature will be measured from the medial longitudinal arch with a thermometer.
  Local skin temperature will be measured with a thermometer from : Right and left lower costal margins, the highest point of the iliac crest (superior side) and the posterior superior iliac spine (inferior side).
Pulse | Eight weeks
  Pulse will be measured with a pulse oximeter attached to the fingertip.
Saturation | Eight weeks
  Saturation will be measured with a pulse oximeter attached to the fingertip.
Blood Pressure | Eight weeks
  The patients' blood pressure will be measured with a sphygmomanometer
The Respiratory Frequency | Eight weeks
  The respiratory frequency value will be obtained by multiplying the number of breaths in and out for thirty seconds by two.
Sit and Reach Test | Eight weeks
  Flexibility will be evaluated with the sit and reach test. Subjects will be asked to sit on the floor to be tested and place their bare feet flat on the test stand. The subject will be asked to lean forward from the body and will extend his/her hands in front of his body as far forward as he can without bending his knees. The farthest point shown by the fingertip will be measured with the help of a tape measure.
Grip Strength | Eight weeks
  Grip Strength is evaluates the strength of the hand muscles used to grasp. In the test procedure, three measurements are made for hand grip strength,and the averages are recorded separately for right and left.
Pittsburgh Sleep Quality Index | Eight weeks
  Pittsburgh sleep quality index, consists of 19 items grouped according to seven component scores. Scores on the seven components are then summed to give a global Pittburgh Sleep Quality İndex score ranging from 0 to 21. Scores between 0 and 4 indicate good sleep quality, scores between 5 and 10 indicate poor quality, and above 10 indicate sleep disturbance.
6-Minute Walk Test | Eight weeks
  The 6-minute walk test measures the maximum distance in meters that a person can walk as fast as possible over a 6-minute period.
Perceived Stress Scale | eight weeks
  Perceived stress scale, is a 10-item that assesses the amount of perceived psychological stress during the past month. Participants evaluate each item on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". A high score indicates a person's perception of stress is high
The Fatigue Severity Scale | Eight weeks
  The fatigue severity scale, evaluates how fatigue affects motivation, exercise, physical functioning, performance of tasks, work, family and social life. It is scored on a 7-point Likert scale. A total score is 9-63 , and a score of 36 and above indicates severe fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem TÜTÜN YÜMİN, Professor, Study Director — Bolu Abant İzzet Baysal University
Locations (1):
- Abant Izzet Baysal University, Bolu, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No